CLINICAL TRIAL: NCT05199558
Title: Improved Characterisation of Eclampsia to Optimise Maternal and Perinatal Outcomes:A Prospective Observational Multicentric Study.
Brief Title: Improved Characterisation of Eclampsia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yousra M. Othman, Principle investigator , assistant lecturer of obstetrics and gynecology, Assiut University, Egypt, Assiut University
Other Study IDs: Prediction of Eclampsia
Record Dates: First submitted 2021-12-31; First posted 2022-01-20 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2021-12

CONDITIONS: Eclampsia Preeclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- eclamptic patients
- preeclamptic patients
- healthy pregnant women of same gestation and parity

SUMMARY:
Eclampsia is a serious pregnancy complication.In our study we aim to characterize the clinical signs and symptoms that occur prior to the onset of eclampsia in a prospectively collected cohort.And Compare these characteristics to women with preeclampsia and healthy normal pregnancies to identify which features represent a unique clinical signature for eclampsia to form a simple predictive algorithm .

DETAILED DESCRIPTION:
Eclampsia is a serious pregnancy complication that occurs when a pregnant woman - or new mother - experiences seizures associated with hypertension. These seizures pose a major risk to the life and the health of mothers and unborn babies. Signs or symptoms of severe preeclampsia are not always present or easy to recognise before a woman develops eclampsia. This is why it can be difficult to tell which women are likely to develop eclampsia before the first seizure occurs. If we can identify the features that are most common and unique to eclampsia, these could be used to develop a tool to help identify the women displaying signs or symptoms that occur prior to the onset of eclamptic seizures. This would mean that treatment to prevent seizures could be targeted to the right women and quickly administered before they become extremely unwell with this life-threatening complication.

Rates of eclampsia are far greater in low to middle income countries , with an estimated 16-69 cases of eclampsia per 10,000 livebirths. Thus, research conducted in LMIC settings allow for the prospective recruitment of a relatively large cohort of women with eclampsia. They are a useful target population to prospectively characterise the signs and symptoms preceding the disease. Such characterisation may yield a unique clinical signature for eclampsia and the development of a predictive algorithm.

ELIGIBILITY:
Inclusion Criteria:

1. Eclampsia:

   * Diagnosed as new onset generalized tonic colonic seizures or coma in pregnant women or women who have recently given birth.
   * Singleton pregnancies.
   * All gestational ages, including post-partum eclampsia
   * Enrolment to the study must occur within 7 days of an eclamptic episode Women must be coherent and able to provide informed consent prior to enrolment
2. Preeclampsia:

   ● Diagnosed as new onset of hypertension (>140 mmHg systolic or > 90 mmHg diastolic) after the 20th week of gestation and the coexistence of one or more of the following new onset conditions:Proteinuria ,Other maternal organ evolvement.
   * Singleton pregnancy.
   * Have not experience an eclamptic episode
3. Normotensive controls:

   * Healthy normotensive pregnant woman recruited from women seeking maternity services during the same or similar period
   * Matched 1:1 for each eclampsia and preeclampsia case
   * Matched by closest gestational age at recruitment to cases and parity

Exclusion Criteria:

* Women with multiple pregnancies.
* Women with seizures attributed to a diagnosis other than eclampsia such as; central nervous system infections, a history of seizures or epilepsy, medications and/or illicit drug use.
* Women unable to provide informed consent

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — pregnant women with preeclampsia\eclampsia.
Study Population: Pregnant women with preeclampsia and eclampsia who will be admitted to Women Health Hospital , Assiut University compared to healthy normotensive pregnant woman recruited from women seeking maternity services during the same or similar period at same gestational age and parity .
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Numbers of clinical features ( symptoms and signs) of eclampsia that can make a predictive model for eclampsia. | 2 years
  estimate the presence or absence of a clinical signature of imminent eclampsia

REFERENCES:
- [Background] Osungbade KO, Ige OK. Public health perspectives of preeclampsia in developing countries: implication for health system strengthening. J Pregnancy. 2011;2011:481095. doi: 10.1155/2011/481095. Epub 2011 Apr 4. PMID 21547090
- [Background] Frias AE Jr, Belfort MA. Post Magpie: how should we be managing severe preeclampsia? Curr Opin Obstet Gynecol. 2003 Dec;15(6):489-95. doi: 10.1097/00001703-200312000-00006. PMID 14624215